CLINICAL TRIAL: NCT06447103
Title: 89Zr-DFO-GmAb PET/CT vs Contrast-Enhanced CT for Detection of Recurrent Clear Cell Renal Cell Carcinoma After Surgery
Brief Title: An Investigational Scan (89Zr-DFO-GmAb PET/CT) Compared to Contrast-Enhanced CT for the Detection of Recurrent Clear Cell Renal Cell Cancer After Surgery Comparing Carbonic Anhydrase IX (CAIX) PET CT to Conventional PET CT for Post-Op Staging in Kidney Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-001576; NCI-2024-01928 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-06-03; First posted 2024-06-06 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Clear Cell Renal Cell Carcinoma; Sarcomatoid Renal Cell Carcinoma; Stage II Renal Cell Cancer; Stage III Renal Cell Cancer; Stage IV Renal Cell Cancer
Keywords: Renal
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (89Zr-DFO-GmAb PET/CT) (Experimental): Patients receive 89Zr-DFO-GmAb IV over 3 minutes on day 0 then undergo whole body PET/CT and SOC diagnostic contrast-enhanced CT scan on day 7. Patients also blood sample collection on study. In addition, patients may undergo bone scan and CT or MRI of the brain on study as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Zirconium Zr 89 Girentuximab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT, PET/CT, and CT of the brain
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI of the brain
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Questionnaire Administration — Ancillary studies
Drug: Zirconium Zr 89 Girentuximab — Given IV
  Other Names: 89Zr-DFO-TFP-girentuximab; 89Zr-girentuximab; 89Zr-TLX250; Zirconium Zr 89 cG250; Zirconium Zr 89-TLX250

SUMMARY:
This phase II trial compares the safety and effectiveness of 89Zr-DFO-GmAb positron emission tomography (PET)/computed tomography (CT) compared to contrast-enhanced CT after surgery in detecting clear cell renal cell cancer that has come back (recurrent). For some patients, the risk of recurrence after surgery remains high. Conventional CT methods, such as contrast-enhanced CT, may not detect small volume or micrometastatic disease. PET/CT with radiotracers, such as 89Zr-DFO-GmAb, may improve detection of tumor cells. Girentuximab (GmAb), a monoclonal antibody, is tagged with zirconium-89, a radioactive atom (which is also known as an isotope). The zirconium-89 (89Zr) isotope is attached to girentuximab with desferrioxamine (DFO) and this combined product is called 89Zr-DFO-girentuximab. 89Zr-DFO-girentuximab attaches itself to a protein on the surface of clear cell renal cell tumor cells called CAIX. PET is an established imaging technique that utilizes small amounts of radioactivity attached to very minimal amounts of tracer, in the case of this research, 89Zr-DFO-GmAb. Because some cancers, including clear cell renal cell cancer, take up 89Zr-DFO-GmAb it can be seen with PET. CT utilizes x-rays that traverse body from the outside. CT images provide an exact outline of organs and potential inflammatory tissue where it occurs in patient's body. Using contrast agents with CT scan to enhance the images (contrast-enhanced CT) is standard of care imaging. 89Zr-DFO-GmAb PET/CT may be safe and effective compared to contrast-enhanced CT in detecting recurrent clear cell renal cell cancer after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the lesion detection rate (i.e., positivity rate per patient) of zirconium Zr 89 girentuximab (89Zr-DFO-GmAb) PET/CT compared to the standard of care diagnostic contrast-enhanced CT alone at 4-12 weeks from surgical resection based on blinded independent central review (BICR).

SECONDARY OBJECTIVES:

I. To establish safety of 89Zr-DFO-GmAb in patients with intermediate-high or high risk imaged in the post-nephrectomy or metastasectomy setting.

II. To compare the positive predictive value (PPV) of 89Zr-DFO-GmAb PET/CT in patients with available lesion validation by 1) histopathology (biopsy/resection), 2) evidence of growth under surveillance or 3) reduction of size under treatment, and 4) unequivocal confirmation of malignancy on a different imaging modality.

III. To assess the recurrence-free survival of individuals with/without evidence of disease based on 89Zr-DFO-GmAb PET/CT staging results (PET/CT designated M1 versus [vs] M0).

EXPLORATORY OBJECTIVES:

I. Correlate level of histological CAIX expression (H Score) from the primary tumor to 89Zr-TLX250 standardized uptake values (SUVs) in patients with visualized disease on 89Zr-DFO-GmAb PET/CT.

II. To identify the standardized uptake value (SUV) cut-off for 89Zr-DFO-GmAb suitable for the detection of metastatic lesions in the postoperative setting.

III. To evaluate the performance of established prognostic transcriptomic classifiers (from the nephrectomy specimen) on disease-free survival.

IV. To evaluate if circulating tumor DNA (ctDNA) for the detection of molecular residual disease (MRD) correlates with the presence of active disease seen on 89Zr-DFO-GmAb PET/CT or predicts disease-free survival.

OUTLINE:

Patients receive 89Zr-DFO-GmAb intravenously (IV) over 3 minutes on day 0 then undergo whole body PET/CT and standard of care (SOC) diagnostic contrast-enhanced CT scan on day 7. Patients also blood sample collection on study. In addition, patients may undergo bone scan and CT or magnetic resonance imaging (MRI) of the brain on study as clinically indicated.

After completion of study intervention, patients are followed up at 8, 16 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Histologically confirmed clear cell renal cell carcinoma (RCC) (ccRCC) (based on partial/radical nephrectomy/metastasectomy)

  * For tumors with extensive sarcomatoid features, if there is evidence of areas of clear cell and high CAIX expression throughout the tumor on immunohistochemistry, they will be allowed on study
* Subjects must have undergone definitive treatment of their primary tumor (partial/radical nephrectomy) +/- resection of metastatic disease to no evidence of disease (NED) with a prior nephrectomy < 2 years)
* Surgery must have been performed between 4-16 weeks at the time of planned imaging
* Subjects are considered to have a high risk of recurrence based on the following criteria:

  * Intermediate-high risk ccRCC:

    * pathologic tumor stage 2 (pT2), grade 4, or sarcomatoid, N0, M0
    * pathologic tumor stage 3 (pT3), any grade, N0, M0
  * High risk ccRCC:

    * pathologic tumor stage 4 (pT4), any grade, N0, M0
    * pT any stage, any grade, number of positive nodes (pN+), M0
  * M1 now NED: pathologically-confirmed ccRCC, undergoing a resection of a solitary, isolated soft tissue metastasis within two years from initial nephrectomy
* Negative serum pregnancy tests in female patients of childbearing potential. (Women of child bearing potential [WOCBP] require a negative pregnancy test within 24 hours (urine) prior to receiving investigational product)
* Consent to practice double-barrier contraception until a minimum of 42 days after 89Zr-DFO-GmAb administration
* Individual must be able to remain still and lie flat for duration of the diagnostic imaging procedure (less than 1 hour)

Exclusion Criteria:

* Inability to provide written informed consent
* Any evidence of residual disease or known metastasis at the time of planned 89Zr-DFO-GmAb administration
* Prior post-operative imaging for confirmation of disease status
* An untreated non-renal malignancy with the following exceptions:

  * Low risk prostate cancer on active surveillance (National Comprehensive Cancer Network [NCCN] very low/low risk)
  * Non-melanoma skin cancer
* Any prior treated malignancy meeting the following characteristics:

  * Treated stage I or II cancer from which the patient is currently in complete remission
  * A stage III cancer from which the patient is progressing or has been disease-free for and has required active treatment (e.g. adjuvant or maintenance therapy) within the past 3 years prior to enrollment
  * A hematologic malignancy from which the patient is currently in complete remission
* Contraindication to the use of iodinated contrast-enhanced CT agents, based on:

  * Severe allergy (for which pre-medication cannot limit adverse reactions) or
  * Estimated glomerular filtration rate (GFR) ≤ 30 ml/min/1.73m^2
* Prior use of systemic therapy treatment for kidney cancer (PD-1, PD-L1, tyrosine kinase or TOR inhibitor) or radiotherapy within 4 weeks of enrollment
* Exposure to experimental diagnostic or therapeutic drug within 14 days from date of planned administration
* Women who are pregnant or breastfeeding
* Known hypersensitivity to girentuximab
* Known inability to remain still and lie flat imaging procedure (about 30 minutes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Lesion detection rate | Up to 16 weeks from surgical resection
  Patients will be treated as binary categorization as follows: (i) Patients who have ≥ 1 lesion confirmed to be recurrent disease will be designated positive (recurrence). (ii) Patients with no lesions detected will be designated negative (no recurrence). The analysis of the primary objective will utilize McNemar's test to compare the detection rate between the imaging techniques.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to day 14
  The total number of AEs will be summarized with grade and attribution. The total number of significant AEs will be summarized with attribution if present. AEs will be descriptive in nature and only counts and percentage will be reported.
Positive predictive value (PPV) | Up to 2 years
  Will compare PPV of 89Zr-DFO-GmAb PET/CT in subjects designated as having a suspicious lesion on the BICR PET/CT evaluation, will review follow up for available lesion validation by 1) histopathology (biopsy/resection), 2) evidence of growth under surveillance or 3) reduction of size under treatment, and 4) unequivocal confirmation of malignancy on a different imaging modality. As there are no firm estimates to the number of lesions that will be designated as suspicious, there are no planned statistical analyses planned. Would present the total number of cases and the frequency of validation with the 95% confidence interval.
Recurrence-free survival | Up to 2 years
  Recurrence-free survival will be calculated using the Kaplan-Meier Method with date and evidence of recurrence based on either clinical annotation by the treating physician or documentation of recurrence by diagnostic imaging or histopathology. Analysis will be descriptive and provide an estimated 2-year recurrence-free survival with 95% confidence interval. A Log-rank test will compare the differences in recurrence-free survival between groups.
Change in management and perceived clinical utility of the unblinded read/report of positron emission tomography/ computed tomography (PET/CT) | At baseline and up to 2 years
  Questionnaires using Likert scores will be used to determine changes. Analysis will be descriptive.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Shuch, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States